CLINICAL TRIAL: NCT00819975
Title: Differential Effects of Milk Proteins on Postprandial Lipemia in Response to a Fat-Rich Meal in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Obesity Research Centre (Other); Nordic Centre of Excellence (Other); Arla Foods (Industry)
Responsible Party: Kjeld Hermansen, Professor, Chief Physician, MD, Dr.Med.Sci, Department of Endocrinology and Metabolism, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-PPL (5B) LSM
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Postprandial Lipemia; Type 2 Diabetes
Keywords: Casein; Whey; postprandial; Triglyceride; Free fatty acids; Retinyl palmitate; Incretins; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caseins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Casein (Active Comparator)
  Interventions: Dietary Supplement: Casein
- Whey Isolate (Active Comparator)
  Interventions: Dietary Supplement: Whey Isolate
- Whey Hydrolysate (Active Comparator)
  Interventions: Dietary Supplement: Whey Hydrolysate
- Alphalact-Albumin (Active Comparator)
  Interventions: Dietary Supplement: Alphalact-Albumin

INTERVENTIONS:
Dietary Supplement: Casein
  Arms: Casein
Dietary Supplement: Whey Isolate
  Arms: Whey Isolate
Dietary Supplement: Whey Hydrolysate
  Arms: Whey Hydrolysate
Dietary Supplement: Alphalact-Albumin
  Arms: Alphalact-Albumin

SUMMARY:
Enhanced and prolonged postprandial triglyceride responses involve increased cardiovascular risk in type 2 diabetes. It has been demonstrated that dietary fat and carbohydrates profoundly influence postprandial hypertriglyceridemia in type 2 diabetes, whereas little information exists about the effect of proteins.

The purpose of this study is to compare the effects of the milk proteins casein, Whey Isolate, Whey Hydrolysate, and Alphalact-Albumin on postprandial lipid and incretin responses to a high-fat meal in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes

Exclusion Criteria:

* Liver-, Kidney- and/or Heart Disease
* Serious Hypertension (160/110 mmHg)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Triglyceride levels | 0h- 2h- 4h- 6h- 7h- 8h postprandial

SECONDARY OUTCOMES:
Incretin levels | 0h- 0.5h- 1h- 2h- 4h- 6h- 8h postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Professor, MD, Principal Investigator — Department of Endocrinology and Metabolism
Locations (1):
- Department of Clinical Nutrition, Aarhus, Denmark